CLINICAL TRIAL: NCT04078594
Title: Stepped-wedge Cluster Randomized Controlled Trial of Electronic Early Notification of Sepsis in Hospitalized Ward Patients (SCREEN)
Brief Title: Electronic Early Notification of Sepsis in Hospitalized Ward Patients
Acronym: SCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: King Abdulaziz Medical City, Jeddah (Unknown); Prince Mohammed Bin Abdul Aziz Hospital - AlMadinah (Unknown); King Abdulaziz Hospital, Al Ahsa (Unknown); Imam Abdulrahman Al Faisal Hospital - Dammam (Unknown)
Responsible Party: Principal Investigator, Dr Yaseen Arabi, Chairman intensive care unit, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC18/112
Record Dates: First submitted 2019-01-17; First posted 2019-09-06 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2021-08

CONDITIONS: Sepsis
Keywords: sepsis; ward patients; Screening; qSOFA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Stepped-wedge Cluster Randomized Controlled Trial
Masking Description: The electronic alert will be masked on the control wards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental wards (Experimental): Active sepsis e-alert
  Interventions: Other: sepsis e-alert
- Contol wards (No Intervention): Masked sepsis e-alert.
  The wards will have masked sepsis e-alert.

INTERVENTIONS:
Other: sepsis e-alert — At 2-each month interval, the e-alert will be activated in five new randomly selected wards, until all wards eventually will have active alert
  Arms: Experimental wards

SUMMARY:
Screening for sepsis has been recommended by the Surviving Sepsis Campaign Clinical Practice Guidelines to facilitate early identification and early management of sepsis. However, the optimal tool remains unknown.The objective of this trial is to examine the effect of an electronic sepsis alert tool on reducing hospital mortailty in patients admitted to medical-surgical-oncology wards.

DETAILED DESCRIPTION:
The study aims to examine the effect of screening for sepsis using an electronic sepsis alert versus no alert in hospitalized patients admitted to wards using an active sepsis alert system compared with wards with no active (masked) sepsis alert system on hospital mortality by day 90.

The wards will be randomized in a stepped-wedge cluster fashion.

ELIGIBILITY:
Ward level inclusion and exclusion criteria

Inclusion Criteria:

1. Inpatient wards, defined as wards used to manage inpatients, in the five Ministry of National Guard Health Affairs (MNGHA) hospitals, Kingdom of Saudi Arabia

Exclusion Criteria:

1. Cardiology, transplant, pediatric, obstetric wards
2. Intensive Care Units and Emergency Department
3. Operating rooms
4. Outpatients
5. Day care wards, endoscopy, outpatient procedure areas, hemodialysis units.

Patient level inclusion and exclusion criteria

Inclusion Criteria:

1. Aged 14 years or older
2. Checked in as inpatient status to one of the study ward

Exclusion Criteria:

1. No commitment for full life support on the time of arrival to the study ward

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65250 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
All-cause hospital mortality by day 90 | 90 Day
  Percentage of all-cause hospital mortality

SECONDARY OUTCOMES:
Hospital length of stay | 90 Day
  Censored at 90 days
Transfer to ICU | 90 Day
  ICU admission within 90 days
ICU-free days | 90 Day
  In the first 90 days
Critical care response team activation | 90 Day
  Critical care response team activation within 90 days
Cardiac arrest | 90 Day
  Cardiac arrest within 90 days
The need for mechanical ventilation, vasopressor therapy, and incident renal replacement therapy | 90 Day
  Within 90 days
Antibiotic-free days | 90 Day
  Antibiotic-free days within 90 days
The acquisition of MDROs | 90 Day
  The percentage of patients with MDROs within 90 days
Clostridium difficile infection | 90 Day
  The percentage of patients with clostridium difficile infection within 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Department, King Abdulaziz Medical City, National Guard Health Affairs, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arabi YM, Alsaawi A, Alzahrani M, Al Khathaami AM, AlHazme RH, Al Mutrafy A, Al Qarni A, Vishwakarma RK, Al Anazi R, Al Qasim E, Abdukahil SA, Al-Rabeah FK, Al Ghamdi H, Alatassi A, Al-Dorzi HM, Al-Hameed F, Babakr R, Alghamdi AA, Bin Salih S, Alharbi A, AlKatheri ME, Mustafa H, Al-Qahtani S, Al Qahtani S, Alselaim N, Tashkandi N, Alyami AH, Alyousef Z, AlDibasi O, Al-Qahtani AH, Aldawood A, Caswell A, Al Ayadhi N, Al Rehaili H, Al Arfaj A, Al Mubarak H, Alwasaidi T, Zahrani S, Alalawi Y, Alhadab A, Nasser T, Omer T, Al Johani SM, Alajlan A, Sadat M, Alzunitan M, Al Mohrij S; SCREEN Trial Group and the Saudi Critical Care Trials Group. Electronic Sepsis Screening Among Patients Admitted to Hospital Wards: A Stepped-Wedge Cluster Randomized Trial. JAMA. 2025 Mar 4;333(9):763-773. doi: 10.1001/jama.2024.25982. PMID 39658862
- [Derived] Arabi YM, Vishwakarma RK, Al-Dorzi HM, Al Qasim E, Abdukahil SA, Al-Rabeah FK, Al Ghamdi H, Al Ghamdi E; SCREEN Trial Group. Statistical analysis plan for the Steppedwedge Cluster Randomized trial of Electronic Early Notification of sepsis in hospitalized ward patients (SCREEN). Trials. 2021 Nov 22;22(1):828. doi: 10.1186/s13063-021-05788-3. PMID 34809672
- [Derived] Arabi YM, Alsaawi A, Al Zahrani M, Al Khathaami AM, AlHazme RH, Al Mutrafy A, Al Qarni A, Al Shouabi A, Al Qasim E, Abdukahil SA, Al-Rabeah FK, Al Ghamdi H, Al Ghamdi E, Alansari M, Abuelgasim KA, Alatassi A, Alchin J, Al-Dorzi HM, Ghamdi AA, Al-Hameed F, Alharbi A, Hussein M, Jastaniah W, AlKatheri ME, AlMarhabi H, Mustafa HT, Jones J, Al-Qahtani S, Qahtani S, Qureshi AS, Salih SB, Alselaim N, Tashkandi N, Vishwakarma RK, AlWafi E, Alyami AH, Alyousef Z; SCREEN Trial Group. Electronic early notification of sepsis in hospitalized ward patients: a study protocol for a stepped-wedge cluster randomized controlled trial. Trials. 2021 Oct 11;22(1):695. doi: 10.1186/s13063-021-05562-5. PMID 34635151